CLINICAL TRIAL: NCT07211737
Title: (INCITE-ON) Phase I Study of i15.NKG2D.Zeta-NK Cell Conditioning in the Tumor Micro-environment in Combination With C7R.GD2.CAR-T for the Treatment of Patients With Relapsed or Refractory Osteosarcoma or Neuroblastoma
Brief Title: NKG2D.Zeta-NK Cell Conditioning With C7R.GD2.CAR-T Cells for Patients With Relapsed or Refractory Osteosarcoma or Neuroblastoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Robin Parihar, MD, PhD, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-55743 INCITE-ON
Record Dates: First submitted 2025-09-04; First posted 2025-10-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Relapsed Neuroblastoma; Refractory Neuroblastoma; Relapsed Osteosarcoma; Refractory Osteosarcoma
Keywords: Gene Therapy; CAR T cells; Neuroblastoma; Osteosarcoma; Immunotherapy; chimeric antigen receptor; NK Cell
MeSH Terms: conditions — Neuroblastoma; Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- i15.NKG2D.zeta NK cells and C7R.GD2.CARTs cells (Experimental): Three dose levels will be evaluated. This is a dose escalating trial which will infuse doses of i15.NKG2D.zeta NK cells followed by a fixed dose of C7R.GD2.CAR T cells 5 days later.
  Interventions: Genetic: i15.NKG2D.zeta NK cells and C7R.GD2.CARTs cells

INTERVENTIONS:
Genetic: i15.NKG2D.zeta NK cells and C7R.GD2.CARTs cells — Dose Level 1: 3 x 10^8/m^2 of i15.NKG2D.zeta NK cells and 3 x 10^7/m^2 of C7R.GD2.CAR T cells given 5 days later.
Genetic: i15.NKG2D.zeta NK cells and C7R.GD2.CARTs cells — Dose Level 2: 6 x 10^8/m^2 of i15.NKG2D.zeta NK cells and 3 x 10^7 cells/m^2 of C7R.GD2.CAR T cells given 5 days later.
Genetic: i15.NKG2D.zeta NK cells and C7R.GD2.CARTs cells — Dose Level 3: 12 x 10^8/m^2 of i15.NKG2D.zeta NK cells and 3 x 10^7 cells/m^2 of C7R.GD2.CAR T cells given 5 days later.

SUMMARY:
The purpose of this study is to find the largest safe dose of i15.NKG2D.zeta-NK cells in combination with C7R.GD2.CAR-T cells, and additionally to evaluate how long they can be detected in patients' blood and what affect they have on patients' cancer.

Patients eligible for this study have neuroblastoma or osteosarcoma that expresses a substance on the cancer cells called GD2. This cancer has either come back after treatment or did not respond to the standard or other investigational treatments or therapies used to treat it. There is no standard treatment for these types of advanced cancers at this time. This is a gene transfer research study using special immune cells called NK cells and T cells. NK cells and T cells are types of white blood cell that help the body fight infection.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: NK cells and T cells. T cells are special infection-fighting blood cells that can kill cells infected with viruses and tumor cells. NK cells, another kind of infection-fighting cell, can recognize a wide range of cells in distress, including tumor cells and cells that help protect tumor cells in the cancer environment. Both NK cells and T cells have been used individually to treat patients with cancers. They have shown promise, but have not been strong enough individually to cure most patients.

Investigators have found from previous research that we can put a new gene into T cells that will make them recognize GD2, a substance found on almost all neuroblastoma and osteosarcoma cells. We can also put a new gene into NK cells that help them fight the tumor environment. Investigators know that T cells and NK cells need substances called cytokines to survive but the cells do not get enough cytokines after infusion into the body; therefore, the investigators have added the genes C7R and IL15 into the T and NK cells, respectively, to give each cell a constant supply of cytokine that helps them to survive longer.

The C7R.GD2.CAR-T cells and i15.NKG2D.zeta-NK cells are investigational products not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
To make the T cells, the investigators will take patient's blood and stimulate it with growth factors that make T cells grow. Investigators will use a retrovirus to insert the GD2-targeting chimeric antigen receptor (CAR) into the T cells. To make NK cells, investigators will take blood from healthy donors and stimulate them with growth factors that make NK cells grow. Investigators will also use a retrovirus to insert the tumor environment-targeting NK receptor, called NKG2D.zeta, into the NK cells.

The cells generated will be frozen and stored to give back to the patient. Because patients will have received cells with a new gene in them, patients will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

Patients will be assigned a dose of i15.NKG2D.zeta-NK cells. The assigned dose of cells is based on body weight and height.

In this study, patients will receive the i15.NKG2D.zeta-NK and C7R.GD2.CAR-T cells. On Day -5, the patient will be given an injection of i15.NKG2D.zeta-NK cells into the vein through an IV line at the assigned dose. Before receiving the NK cell infusion, the patient may be given a dose of Benadryl (diphenhydramine) and Tylenol (acetaminophen). The infusion will take between 1 to 10 minutes. Investigators will then monitor the patient in the clinic for about 3 hours. The study was designed to not give doses of lymphodepletion chemotherapy prior to the i15.NKG2D.zeta-NK and C7R.GD2.CAR-T cells. However, some patients may need to receive lymphodepletion chemotherapy prior to the NK cell infusion, based on preliminary study results.

This will be followed by an injection of C7R.GD2.CAR-T cells on Day 0. Before receiving the infusion, the patient may be given doses of Benadryl (diphenhydramine) and Tylenol (acetaminophen). The infusion will take between 1 to 10 minutes. Investigators will monitor the patient in the clinic for about 3 hours. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital. The patient may need to stay in Houston for up to 4 weeks after the infusion so we can monitor for side effects.

The patient will have follow-up visits after the T cell infusion at day -3, day +3, weeks 1, 2, 3, 4, and 8, then at months 3, 6, 9, an d 12, and then twice a year for the next 4 years and annually for the next 10 years. The patient will also have scheduled disease evaluations after the T cell injection at week 6 and then as clinically needed.

Medical test before treatment--

Before being treated, the patient will receive a series of standard medical tests:

* Physical exam
* Blood tests to measure blood cells, kidney and liver function
* Measurements of the tumor by routine imaging studies and/or bone marrow evaluation. We will use the imaging studies that have been used in the past to best assess the tumor: Computed Tomography (CT) scan, Magnetic Resonance Imaging (MRI), Position Emission Tomography (PET/CT), Bone Scan, and/or MIBG scan.
* Pulmonary Function Tests (PFT) to see how well the patient's lungs are working.

Medical tests during and after treatment--

The patient will receive standard medical tests when they are getting the infusions and afterwards:

* Physical exams
* Blood tests to measure blood cells, kidney and liver function
* Measurements of the tumor by routine imaging studies and/or bone marrow evaluation 6 weeks after the infusion (if the bone marrow showed tumor before the infusion).

To learn more about the way the i15.NKG2D.zeta-NK cells and C7R.GD2.CAR-T cells are working and how long they last in the body, an extra amount of blood will be obtained on the day of the NK-cell infusion and the T-cell infusion and at the end of the NK-cell and T-cell infusions, 1, 2, 3, 4, and 8 weeks after the T-cell infusion and every 3 months for the 1st year, every 6 months for the next 4 years and annually for the next 10 years. The amount of blood taken will be based on the patient's weight with up to a maximum of 60 mL (12 teaspoons) of blood to be obtained at any one time. For children, the total amount of blood drawn will not be more than 3 mL (less than 1 teaspoon) per 1 kg of body weight on any one day. This volume is considered safe, but may be decreased if patient is anemic (has a low red blood cell count).

During the time points listed above, if the i15.NKG2D.zeta-NK cells or C7R.GD2.CAR-T cells are found in the patient's blood at a certain amount, an extra 5 mL (about 1 teaspoon) of blood may need to be collected for additional testing.

If the patient has a procedure where tumor samples are obtained, like a repeat bone marrow evaluation or tumor biopsy, the investigators will request a sample to be used for research purposes.

The patient will receive supportive care for any acute or chronic toxicities, including blood components or antibiotics, and other intervention as medically appropriate.

ELIGIBILITY:
PROCUREMENT INCLUSION:

1. Patients with Neuroblastoma that have persistent disease after standard treatment or have relapsed/refractory disease.

   Or

   Patients with Osteosarcoma that have persistent disease after standard treatment or have relapsed/refractory disease.
2. Karnofsky/Lansky score of 60% or greater.
3. Informed consent and assent (as applicable) obtained from parent/guardian and child.
4. Greater than 1 year of age.

PROCUREMENT EXCLUSION:

1. History of hypersensitivity to murine protein-containing products.
2. Known presence of Human Anti-Mouse Antibodies (HAMA).
3. Active autoimmune disease (requiring immunosuppressive treatment in the past 6 months).
4. Primary brain tumor or known brain metastases (on evaluation by MIBG and/or PET if applicable, CT/MRI/LP not required).

TREATMENT INCLUSION:

1. Patients with Neuroblastoma that have persistent disease after standard treatment or have relapsed/refractory disease.

   Or

   Patients with Osteosarcoma that have persistent disease after standard treatment or have relapsed/refractory disease.
2. Karnofsky/Lansky score of 50% or greater
3. Pulse Ox greater than or equal to 90% on room air
4. AST less than 5 times upper limit of normal (less than 10 times upper normal if known with metastatic liver disease)
5. Total bilirubin less than 3 times the upper limit of normal
6. Serum creatinine less than 3 times upper limit of normal
7. Available autologous T-cells with greater than or equal to 20% expressing GD2.CAR
8. Informed consent and assent (as applicable) obtained from parent/guardian and child.
9. Greater than 1 year of age.
10. Recovered from acute toxic effects of all prior chemotherapy and investigational agents before entering this study.

TREATMENT EXCLUSION:

1. History of hypersensitivity to murine protein containing products (patients who have undergone desensitization and successful re-challenge without hypersensitivity reaction are eligible).
2. Known presence of Human Anti-Mouse Antibodies (HAMA).
3. Tumor potentially causing airway obstruction per investigator discretion.
4. Pregnancy or lactation / will not use birth control methods.
5. Currently receiving immunosuppressive drugs (patients on low dose corticosteroids are eligible: less than 0.25 mg/kg/day of prednisone/equivalent).
6. Primary brain tumor or known brain metastases (on evaluation by MIBG and/or PET if applicable, CT/MRI/LP not required).

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2044-04 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rate | 4 weeks post-CAR-T cell infusion
  Proportion of participants with DLTs related to the combination of NK cell and T cell infusions evaluated as per the NCI CTCAE v5.0 criteria
Maximum tolerated dose (MTD) of i15.NKG2D.zeta-NK cells when given in combination with C7R.GD2.CAR-T cells | 4 weeks post CAR-T infusion of the last participant
  The dose level of infused NK cells for which the DLT rate is approximately 0.3

SECONDARY OUTCOMES:
Objective response rate (ORR) | 6 weeks after CAR-T infusion
  Proportion of participants with complete response (CR) or partial response (PR) according to RECIST v1.1 criteria and/or MIBG evaluation (for neuroblastoma)
Cytokine release syndrome (CRS) grade | 4 weeks post CAR-T infusion
  Any grade CRS as evaluated by established clinical CRS Grading Scale

CONTACTS AND LOCATIONS:
Overall Officials: Leander D Timothy, MD, Principal Investigator — Baylor College of Medicine; Shoba A Navai, MD, Principal Investigator — Baylor College of Medicine; Stephanie L Fetzko, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States